CLINICAL TRIAL: NCT01697722
Title: A Retrospective Evaluation of Effectiveness and Cost-effectiveness of Extrafine HFA-BDP Compared With Combination ICS/LABA Therapy in the Management of Asthma in a Representative Population of UK Primary Care Patients
Brief Title: Real-world Effectiveness and Cost-effectiveness of HFA-beclometasone Compared With ICS/LABA Combination Therapy
Acronym: QvarvsCombo
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, David Price, Professor David Price, Research in Real-Life Ltd
Other Study IDs: BA21
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Primary care; Asthma management; Inhaled corticosteroids; Extra-fine hydrofluoroalkane; Long-acting beta-agonist; Fixed-dose combination therapy
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Step-up as FDC ICS/LABA: ICS asthma patients who increased therapy as FDC ICS/LABA (no increase in daily ICS dose).
- Step up as separate therapies: ICS asthma patients who increased therapy as ICS / LABA via separate pMDI and / or BAI inhalers (no increase in daily ICS dose).
  Interventions: Drug: ICS / LABA via separate pMDI and / or BAI inhalers
- Qvar step-up: ICS asthma patients who increased therpy as extra-fine hydrofluoroalkane-beclometasone dipropionate
  Interventions: Drug: Extra-fine hydrofluoroalkane-beclometasone dipropionate

INTERVENTIONS:
Drug: Extra-fine hydrofluoroalkane-beclometasone dipropionate — Increase in the baseline BDP-equivalent dose of inhaled corticosteroid as HFA-BDP via pMDI or BAI
  Other Names: Qvar
  Groups: Qvar step-up
Drug: ICS / LABA via separate pMDI and / or BAI inhalers — A step-up from baseline ICS therapy via the addition of a separate long-acting beta-agonist with no change in baseline ICS drug or dose
  Other Names: ICS+LABA separates
  Groups: Step up as separate therapies

SUMMARY:
This study will compare the effectiveness, cost-effectiveness and direct healthcare costs of asthma management in patients with evidence of persistent asthma following an increase in asthma therapy in the form of either an increased dose of inhaled glucocorticosteroids (ICS) using extrafine hydrofluoroalkane-beclometasone dipropionate (HFA-BDP) via pressurised metered-dose inhaler (pMDI) or breath-actuated inhaler (BAI), or a change to combination ICS plus long-acting bronchodilator (LABA) therapy using fixed combinations (fluticasone propionate / salmeterol [FP/SAL] or budesonide / formoterol [BUD/FOR]) or separate pMDIs and BAIs.

DETAILED DESCRIPTION:
Current asthma guidelines in the UK are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, the patients recruited to asthma RCTs are estimated to represent less than 10% of the United Kingdom's (UK's) asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is therefore a need for more representative RCTs and real-life observational studies to inform existing guidelines and help optimise asthma outcomes.

The fixed combination asthma inhalers, FP/SAL (Seretide) and BUD/FOR (Symbicort) are indicated for use in asthma when adequate asthma control is not achieved with low/medium dose ICS therapy and as-needed (prn) reliever therapy (a short-acting beta-agonist [SABA]). Fixed combination inhalers are also indicated in patients already adequately controlled on separate ICS/LABA therapy. However, emerging trends in asthma prescribing indicate increasing use of add-on therapies (particularly in the form of combination inhalers) in the early stages of asthma therapy, even as first-line therapy.

In practice, there is significant pressure (supported by asthma guidelines) to use the least expensive, effective inhaled therapies available. While the effect of increased use of add-on and combination therapies in terms of patient benefits remains uncertain, the impact on the UK's National Health Service (NHS) treatment costs is unequivocal.

Short, randomised trials of the effectiveness of asthma monotherapies have demonstrated that extrafine HFA-BDP is at least as effective at half the dose as BDP pMDI, and equivalent to same-dose FP pMDI. There is also evidence to suggest that extrafine HFA-BDP optimises deposition in the lung and affords greater tolerance of poor coordination of breathing and inhaler actuation. In addition, one long-term, prospective, randomised, open-labelled trial comparing extrafine HFA-BDP with BDP over the course of one year demonstrated greater improvements in symptom-free days and quality of life in the extrafine HFA-BDP treatment group, at a lower cost per symptom-free day.

The hypothesis for this study, therefore, is that extrafine HFA-BDP may be a suitable, and cost-effective, alternative to combination therapy (as fixed or separate inhalers) in children and adults with evidence of persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 4-60 years:

  * Paediatric cohort (aged 4-11 years), and
  * Adult cohort (aged 12-60 years)
  * Aged 61-80 years and never smoked for an additional elderly cohort;
* Evidence of asthma: i.e. a diagnostic code of asthma or at least 2 asthma prescriptions, including one ICS prescription, at different points in time during the year prior to IPD (the baseline year)
* Be on current asthma therapy: i.e. at least 1 asthma prescription in the year prior to IPD, and at least 1 other asthma prescription during the same period
* Have at least one year of up-to-standard (UTS) baseline data (prior to the IPD) and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

* had a diagnostic read code for chronic obstructive pulmonary disease (COPD) at any time
* had a diagnostic read code for chronic respiratory disease at any time (other than asthma)
* any patients receiving a combination inhaler in addition to their separate ICS inhaler in the baseline year

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care asthma patients who were receiving ICS therapy (any of BDP, extrafine BDP-HFA, BUD or FP as pMDI or BAI) who, at an index prescription date, underwent either:
  (i) an increase in ICS as extrafine HFA-BDP (pMDI or BAI); (ii) a change to combination therapy with a separate LABA pMDI or BAI (no change in drug, device or daily BDP-equivalent dose) (iii) a change to combination therapy via a fixed-combination inhaler (with no increase in daily BDP-equivalent dose).
Sampling Method: Non-Probability Sample
Enrollment: 815377 (Actual)
Dates: Start 1991-01; Primary Completion 2007-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Proxy asthma control | One-year outcome period
  * No recorded hospital attendance for asthma including admission, Accident & Emergency (A&E) attendance, out of hours attendance or Out-Patient Department (OPD) attendance, AND
  * No prescriptions for oral steroid, AND
  * No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics

SECONDARY OUTCOMES:
Success of therapeutic regimen | One-year outcome period
  Defined as the absence of (i) Exacerbation:
  1. Unscheduled hospital admissions / A&E attendance for asthma, OR
  2. Acute use of oral steroids
  AND
  (ii) No consultations, hospital admissions or A&E attendance for LRTI requiring antibiotics
  AND
  (iii) No change in therapeutic regimen:
  1. Increased dose of ICS, and/or
  2. Change in ICS/LABA, and/or
  3. Change in delivery device, and/or
  4. Use of additional therapy as defined by: theophylline, LTRAs, oral beta agonists (or LABAs in patients receiving extrafine HFA-BDP).
Success of therapeutic regimen (sensitivity - independent of cost saving) | One-year outcome period
  Success: defined as the absence of
  (i) Exacerbation:
  1. Unscheduled hospital admissions / A&E attendance for asthma, OR
  2. Acute use of oral steroids
  AND
  (ii) No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics
  AND
  (iii) No change in therapeutic regimen:
  1. Increased dose of ICS, and/or
  2. Use of additional therapy as defined by: theophylline, leukotreine receptor antagonists (LTRAs), oral beta agonists (or LABAs in patients receiving extrafine HFA-BDP).
average SABA daily dose during outcome year | One-year outcome period
  Average daily dose categorised as: 0mcg, >0-100mcg, >100-200mcg, >200-400mcg, >400-800mcg, >800mcg).
Hospitalisations | One-year outcome period
  Mean number of asthma and respiratory-related hospitalisations recorded per patient during the outcome year

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof. MD, Principal Investigator — Company Director; Alison Chisholm, MSc, Study Director — Research Project Director
Locations (1):
- General Practice Research Database, London, London, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma. National Heart, Lung, and Blood Institute, National Institutes of Health, 2007. (Accessed March 2008, at http://www.nhlbi.nih.gov/guidelines/asthma/asthgdln.pdf
- [Background] Aubier M, Wettenger R, Gans SJ. Efficacy of HFA-beclomethasone dipropionate extra-fine aerosol (800 microg day(-1)) versus HFA-fluticasone propionate (1000 microg day(-1)) in patients with asthma. Respir Med. 2001 Mar;95(3):212-20. doi: 10.1053/rmed.2000.1025. PMID 11266239
- [Background] Fairfax A, Hall I, Spelman R. A randomized, double-blind comparison of beclomethasone dipropionate extrafine aerosol and fluticasone propionate. Ann Allergy Asthma Immunol. 2001 May;86(5):575-82. doi: 10.1016/S1081-1206(10)62907-9. PMID 11379810
- [Background] Lasserson TJ, Cates CK, Jones AB, Steele EH, White J. Fluticasone versus HFA-beclomethasone dipropionate for chronic asthma in adults and children. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD005309. doi: 10.1002/14651858.CD005309.pub3. PMID 16625634
- [Background] Gross G, Thompson PJ, Chervinsky P, Vanden Burgt J. Hydrofluoroalkane-134a beclomethasone dipropionate, 400 microg, is as effective as chlorofluorocarbon beclomethasone dipropionate, 800 microg, for the treatment of moderate asthma. Chest. 1999 Feb;115(2):343-51. doi: 10.1378/chest.115.2.343. PMID 10027430
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org